CLINICAL TRIAL: NCT02944474
Title: A Randomised Double-blind, Placebo-controlled, Ascending Multiple Dose Phase 1 Study of CDP923 in Healthy Volunteers to Assess Safety, Tolerability, Pharmacokinetics and Food Effect
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of Lucerastat (CDP923) After Multiple Dosing in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CDP923-002
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Healthy Subjects
Keywords: Pharmacokinetics; Safety
MeSH Terms: interventions — migalastat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (200 mg) (Experimental): Six subjects received 200 mg of lucerastat twice daily for 7 consecutive days in fasting conditions
  Interventions: Drug: Lucerastat
- Cohort 2 (500 mg) (Experimental): Six subjects received 500 mg of lucerastat as a single dose in the morning of Day 1 in fed conditions. After a 5-day washout, they received the same dose twice daily for 7 consecutive days in fasting conditions
  Interventions: Drug: Lucerastat
- Cohort 3 (500 mg) (Experimental): Six subjects received 500 mg of lucerastat twice daily for 7 consecutive days in fasting conditions
  Interventions: Drug: Lucerastat
- Cohort 4 (1000 mg) (Experimental): Six subjects received 1 g of lucerastat for 7 consecutive days in fasting conditions
  Interventions: Drug: Lucerastat
- Placebo cohorts 1 to 4 (Placebo Comparator): Twelve subjects received matched placebo (3 subjects per cohort, except for Cohort 3 where 4 subjects received placebo)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lucerastat — Capsule for oral administration containing lucerastat
  Other Names: OGT-923; ACT-434964; CDP923
  Arms: Cohort 1 (200 mg); Cohort 2 (500 mg); Cohort 3 (500 mg); Cohort 4 (1000 mg)
Drug: Placebo — Placebo capsules matching lucerastat capsules
  Arms: Placebo cohorts 1 to 4

SUMMARY:
The objectives of this study were to evaluate the safety and tolerability of lucerastat and to determine its pharmacokinetic profile after multiple dosing. Also, the potential effect of food on the pharmacokinetics of lucerastat was explored following a single dose of 500 mg.

DETAILED DESCRIPTION:
The subjects were to be enrolled sequentially to three dose groups, starting with the lowest dose level. Subjects could participate in only one Group. Progression to an increased dose of lucerastat was permitted only after review of all data from the previous cohort suggested that it was safe to do so.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Male subjects aged from 18 to 45 years at screening.
* Body weight between 50 and 100 kg and body mass index (BMI) between 18.0 and 29.0 kg/m2 at screening.
* Healthy on the basis of physical examination, cardiovascular assessments and laboratory tests.

Exclusion Criteria:

* History or clinical evidence of any disease or medical / surgical condition or treatment, which may put the subject at risk of participation in the study or may interfere with the absorption, distribution, metabolism or excretion of the study treatments.
* Serious adverse reaction or hypersensitivity to any drug.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2003-12; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Dose proportionality in lucerastat pharmacokinetics assessed by maximum plasma concentration (Cmax) | PK blood samples were collected on Day 7, at pre-dose and at scheduled time points up to 48 hours after the morning dose
  Cmax was used to assess dose proportionality across all dose groups
Dose proportionality in lucerastat pharmacokinetics assessed by area under the concentration-time curve (AUC) | PK blood samples were collected on Day 7, at pre-dose and at scheduled time points up to 48 hours after the morning dose on Day 7
  AUC from time zero to infinity [AUC(0-inf)] was used to assess dose proportionality across all dose groups
Terminal elimination half-life (t1/2) | PK blood samples were collected on Day 7, at pre-dose and at scheduled time points up to 48 hours after the morning dose on Day 7
  t1/2 was calculated from the plasma concentrations-time curves of lucerastat after multiple doses
Food effect on lucerastat pharmacokinetics assessed by Cmax | PK blood samples were collected on Day 1, at pre-dose and at scheduled time points up to 12 hours after the morning dose
  Potential food effect on pharmacokinetic parameters of lucerastat was tested by comparing Cmax in fed vs fasted state in the 500 mg cohort (cohort 2)
Food effect on lucerastat pharmacokinetics assessed by AUC | PK blood samples were collected on Day 1, at pre-dose and at scheduled time points up to 12 hours after the morning dose
  Potential food effect on pharmacokinetic parameters of lucerastat was tested by comparing AUC in fed versus fasted state in the 500 mg cohort (cohort 2)
Number of participants with adverse events (AEs) | From baseline up to Day 14 (end of study)
  An AE was defined as any untoward medical occurrence in a clinical investigation subject, which did not necessarily have a causal relationship with the treatment
Change from baseline in haematology after multiple doses of lucerastat | Up to Day 9
Change from baseline in clinical chemistry after multiple doses of lucerastat | Up to Day 9
Change from baseline in heart rate after multiple doses of lucerastat | Up to Day 9

SECONDARY OUTCOMES:
Change from baseline in haematology after a single dose of lucerastat | At 24 hours post dose
Change from baseline in clinical chemistry after a single dose of lucerastat | At 24 hours post dose
Change from baseline in heart rate after a single dose of lucerastat | At 24 hours post dose
Change from baseline in blood pressure after a single dose of lucerastat | Up to 24 hours post dose
Change from baseline in electrocardiogram (ECG) variables after a single dose of lucerastat | Up to 24 hours post dose
Stool frequency after multiple doses of lucerastat | Every day up to Day 9
Change from baseline in body weight after multiple doses of lucerastat | At Day 9

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- Investigator Site, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guerard N, Morand O, Dingemanse J. Lucerastat, an iminosugar with potential as substrate reduction therapy for glycolipid storage disorders: safety, tolerability, and pharmacokinetics in healthy subjects. Orphanet J Rare Dis. 2017 Jan 14;12(1):9. doi: 10.1186/s13023-017-0565-9. PMID 28088251